CLINICAL TRIAL: NCT03892954
Title: MicroRNAs as Biomarkers of Pain Intensity in Patients With Chronic Fatigue Syndrome (CFS)
Acronym: CFs
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sami Gabr, Principal investigator, King Saud University
Other Study IDs: RRC
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Chronic Fatigue Syndrome (CFS)
Keywords: MicroRNAs; Chronic fatigue syndrome; Pain intensity
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood was collected from all subjects and serum samples were obtained following centrifugation for 1 min. at 1400 rpm, were given a coded study identification number, and were shipped frozen at 20° C for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adolescents with CFS ( n= 100): Participants with CFS who had constant or persisting fatigue lasting 3 months with the severe functional disability to such extent that prevents normal school attendance and also had no drug prescriptions (including hormone contraceptives), any medical or psychiatric disorder that might explain the fatigue were included in this study
- health control ( n=50).: healthy control subjects with no CFS

SUMMARY:
MicroRNAs were shown to play an important role in regulating pain-processing in a wide range of experimental models and clinical pain disorders. Thus, the aim of the present study is to evaluate a set of Micro-RNAs as diagnostic biomarkers of pain intensity in adolescents with chronic fatigue syndrome (CFS) and to correlate with inflammatory markers and pain related comorbidities.

DETAILED DESCRIPTION:
The present study was performed to evaluate a set of Micro-RNAs as diagnostic biomarkers of pain intensity in adolescents with chronic fatigue syndrome (CFS) and to correlate with inflammatory markers and pain related comorbidities. Thus, a total of 150 adolescents aged (12-18 years) were invited to participate in this study. They are classified into two groups; adolescents with CFS (n=100) and healthy control (n=50). RT-PCR and immunoassay analysis were used to estimate miRNAs (miR-558, miR-146a, miR-150, miR-124, and miR-143) and immune-inflammatory markers (IL-6, TNF-α, COX-2) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants with CFS who had constant or persisting fatigue lasting 3 months with the severe functional disability to such extent that prevents normal school attendance and also had no drug prescriptions (including hormone contraceptives), any medical or psychiatric disorder that might explain the fatigue were included in this study.

Exclusion Criteria:

* Participants who had drug prescriptions (including hormone contraceptives), any medical or psychiatric disorder that might explain the fatigue were excluded from this study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 150 adolescents aged (12-18 years) were invited to participate in this study. Based on CFS diagnosis, participants were classified with CFS (n=100) and healthy controls (n=50). adolescents who had constant or persisting fatigue lasting 3 months with the severe functional disability to such extent that prevents normal school attendance and also had no drug prescriptions (including hormone contraceptives), any medical or psychiatric disorder that might explain the fatigue were included in this study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Assessment of pain intensity | 3-4 weeks
  A pre-validated modified Brief Pain Inventory (BPI) was performed to measure pain scores among both subjects with CFS and healthy controls.The BPI includes four ratings of pain intensity (items 3-7), and seven other ratings on the impact of pain. Intensity is recorded on numerical scales from zero (no pain) to ten (pain as bad as you can imagine). Also, intensity is rated at the time of completing the questionnaires (pain now) as well as its worst, least, and average over the past day or week. The BPI also records the location of the pain on a diagram of a human figure. Patients are also asked to select words that best describe their pain and to indicate the extent and duration of pain relief obtained from analgesics.
Assessment of cyclooxygenase 2 protein (COX-2), tumor necrosis factor (TNF-α) and interleukin-6 (IL-6) as physiological pain regulators | 3-4 weeks
  For all participants, cyclooxygenase 2 protein (COX-2), tumor necrosis factor (TNF-α) and interleukin-6 (IL-6) were estimated in serum samples of CFS and control subjects

SECONDARY OUTCOMES:
Assessment of the levels of Isolated miRNAs in the serum samples. | 8 weeks
  RT-PCR techniques were used to estimate the levels of mi-RNAs in serum samples of CFS and control subjects